CLINICAL TRIAL: NCT03667027
Title: Diaphragm Structure and Pathobiology in Patients Being Bridged to Lung Transplant
Acronym: DIASPORA
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Other Study IDs: 18-5660
Record Dates: First submitted 2018-08-31; First posted 2018-09-12 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Diaphragm Injury; Respiratory Failure; Mechanical Ventilation Complication
Keywords: Diaphragm Dysfunction; Acute Respiratory Failure; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Diaphragm tissue Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients undergoing LTx with respiratory failure (cases): Patients are receiving a respiratory support modality (mechanical ventilation and/or extracorporeal life support) as a bridge to lung transplantation (LTx).
  Interventions: Device: Respiratory support
- Patients undergoing LTx without prior respiratory support: Patients undergoing lung transplantation but do not require prior bridging respiratory support.
- Elective thoracic surgical patients: Patients undergoing elective thoracic surgery for planned lung or esophageal resection.

INTERVENTIONS:
Device: Respiratory support — Mechanical ventilation or extracorporeal life support
  Groups: Patients undergoing LTx with respiratory failure (cases)

SUMMARY:
This study is designed to characterize the changes in diaphragm structure, function and biology during bridging to lung transplant by mechanical ventilation or extracorporeal life support.

DETAILED DESCRIPTION:
Mechanical ventilation has been linked to diaphragm injury and dysfunction. During mechanical ventilation, the amount of breathing work done by the diaphragm is unpredictable: the diaphragm could be completely rested, or it could be overworked. Either of these possibilities may cause injury to the diaphragm. Patients with an injured and dysfunctional diaphragm have greater difficulty weaning from mechanical ventilation - they become too weak to breathe. However, little is known about the relationship between changes in the diaphragm and the histological (structure of cells and tissue) basis of these changes. The investigators have developed a new technique employing beside ultrasound to measure diaphragm thickness. This allows them to observe changes in diaphragm muscle structure and function.

The goal of the study is to determine whether different forms of respiratory support (mechanical ventilation vs extracorporeal life support) lead to different degrees of diaphragm injury and to compare changes in the diaphragm seen on ultrasound to changes in the diaphragm tissues under a microscope. This will help the investigators to confirm the best way to avoid diaphragm injury and to understanding the meaning of diaphragm ultrasound images.

ELIGIBILITY:
Inclusion Criteria (Cases):

* Receiving a respiratory support modality as a bridge to lung transplantation
* Formally listed for transplantation

Inclusion Criteria (Control Group 1):

- Undergoing lung transplantation for either obstructive or restrictive lung disease

Inclusion Criteria (Control Group 2):

- Undergoing elective thoracic surgery without any prior history of chronic pulmonary parenchymal disease

Exclusion Criteria (Cases and Controls):

* Previously diagnosed with neuromuscular disorder
* Received invasive mechanical ventilation for >48 hours in the preceding four weeks
* Thoracic cage deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute respiratory failure awaiting lung transplantation who are being bridged to lung transplantation either by mechanical ventilation or extracorporeal life support.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference in diaphragm thickness and thickening fraction in patients using MV and patients using ECLS | Change from baseline diaphragm thickness and thickening fraction at 7 days after lung transplant
  Diaphragm thickness and injury score will be tested for an interaction between the bridging modality (MV vs. ECLS) and the duration of exposure to the modality on the degree of diaphragm injury and atrophy

SECONDARY OUTCOMES:
Correlate changes in diaphragm thickness and histological features of diaphragm dysfunction | Assessed immediately after transplantation
  Histological features to be assessed are: myofibril cross-sectional area, muscle fiber type, presence of cellular infiltrates, myofiber necrosis and regeneration, autophagy and fibro-fatty infiltration
Biomarkers for diaphragm dysfunction | Assessed immediately before transplantation
  Biomarkers to be assessed are: skeletal troponin-I and markers of systemic inflammation (IL-1, IL-6, Tumor Necrosis Factor (TNF)-alpha)

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No